CLINICAL TRIAL: NCT00020670
Title: A Phase I Study of Vaccination With Autologous CD40-Activated Acute Lymphoblastic Leukemia Cells
Brief Title: Vaccine Therapy in Treating Patients With Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicholas Haining, MD, Haining, Nicholas MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-053; P01CA068484 (NIH); P30CA006516 (NIH); DFCI-00053; NCI-H01-0074
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — FANG vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD40 Cell Vaccination (Experimental): Patients will undergo tumor cell collection followed by vaccine preparation and then vaccination. Autologous acute lymphoblastic leukemia (ALL) cells are harvested, cultured with CD40 ligand, pulsed with keyhole limpet hemocyanin (KLH), and then irradiated to produce the vaccine. Patients receive either 1 x 10^7 or 1 x 10^8 CD40 cells/vaccination depending on the number of tumor cells obtained. Vaccinations are administered every two weeks as outpatient therapy. Evaluable patients receive the course of at least 4 vaccinations at weeks 0, 2, 4, 6. Patients may continue receiving vaccinations every 2 weeks if chemotherapy is not required for symptomatic disease.
  Interventions: Biological: CD 40

INTERVENTIONS:
Biological: CD 40
  Other Names: Autologous tumor cell vaccine

SUMMARY:
The prognosis for children and adults with acute lymphoblastic leukemia (ALL) has improved significantly over the years. Nevertheless, patients who experience disease relapse or induction failure along with patients having unfavorable genetics [t(4;11) or t(9;22)] have dismal prognosis. For these patients, novel therapeutic approaches such as immunotherapy are needed. In this clinical trial, investigators evaluate whether it is feasible to make a vaccine from leukemia cells and whether this vaccine enables direct immunity against cancer cells in patients.

DETAILED DESCRIPTION:
OBJECTIVES Primary

* To determine feasibility of generating a cellular vaccine composed of CD40-activated autologous ALL cells
* To determine feasibility of vaccine administration according to the proposed schedule
* To determine toxicity of vaccination with CD40-activated autologous ALL cells

Secondary

* To assess ALL-specific immunity following vaccination
* To assess the generation of immunity to control antigens
* To develop preliminary information on effect vaccination on tumor response

ELIGIBILITY:
Inclusion Criteria

* B-cell acute lymphoblastic leukemia
* Disease involving at least 30% of bone marrow or circulating blasts
* In first relapse with at least 1 of the following high-risk features:

  * Age under 1 year at diagnosis
  * Age over 18 years at diagnosis
  * t(9;22)
  * Occurrence of first relapse less than 18 months after diagnosis
  * In second relapse or beyond
  * Refractory disease
* Successful generation of adequate CD40 ligand-activated autologous tumor cell vaccine
* Less than 1 year since tumor cell collection
* Patients in first relapse or beyond must be ineligible for or have declined allogeneic bone marrow transplantation in order to receive study vaccine
* Patients need not be in complete remission to receive study vaccine
* Patients may have received an allogeneic hematopoetic stem cell transplant in the past
* No chemotherapy, radiotherapy, immunotherapy or immunosuppressive treatment or within 3 weeks of vaccination
* Adequate hepatic function as defined by: Bilirubin < 2x normal; AST < 3x normal; ALT < 6x normal
* Adequate renal function defined by: Creatinine < 2x normal
* <1 year since tumor cell collection

Exclusion Criteria

* Concurrent treatment as part of another therapeutic research protocol
* Pregnancy or nursing mothers
* Clinically significant pulmonary or cardiac disease
* Clinically significant autoimmune disease
* Documented infection that is active and/or not responding to therapy
* Evidence of HIV infection or known positive HIV serology
* Lansky performance scale (if <18yo) <60%, Karnofsky performance scale (if >18yo) >60%
* Once vaccination course has started: patients may not receive chemotherapy, radiotherapy, immunotherapy or immunosuppressive treatment, hematopoetic growth factors. However between tumor cell collection and vaccine administration, patients may receive non-protocol chemotherapy.

********************************************NOTE***************************************************

It is anticipated that there will be a number of patients at first relapse who are eligible for tumor cell collection and vaccine preparation but who are not eligible to receive the vaccination course. These patients will be evaluable for Objective 3.1.1 (feasibility of vaccine preparation). Patients at first relapse who are eligible for vaccine preparation but not administration should instead be treated with standard salvage regimens which may include allogeneic bone marrow transplantation according to the judgement of their primary oncologist. However, these patients represent a population at extremely high risk for progression of their disease following salvage therapy. Many of these patients will therefore be likely to fulfill eligibility criteria for vaccination in the future (i.e.

should they relapse again, or fail to enter 2nd complete remission). The majority of those patients who relapse for a second time will do so within 1 year. Those patients who become eligible for vaccination because of 2nd relapse within 1 year of tumor cell collection will receive the original vaccine and will not have further vaccine made from tumor cells collected at the time of 2nd relapse. Given the proliferative thrust of the disease in many patients, it will be advantageous to have vaccines already prepared for these patients to reduce the amount of time from 2nd relapse to vaccination.***

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2001-02-20 (Actual); Primary Completion 2003-04-01 (Actual); Study Completion 2003-07-01 (Actual)

PRIMARY OUTCOMES:
Rate Of Successful Vaccine Preparation | 6 weeks
  Vaccine preparation is a success if an adequate number of CD40 activated cells (at least 1 x 10^8 cells) can be generated.

CONTACTS AND LOCATIONS:
Overall Officials: W. Nicholas Haining, BM, BCh, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No